CLINICAL TRIAL: NCT04628351
Title: The Effect of Structured Bladder Training Program on Lower Urinary System Symptoms and Quality of Life After Radical Prostatectomy
Brief Title: Bladder Training in Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, RN, PHD, Asst Prof, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19/37
Record Dates: First submitted 2020-11-07; First posted 2020-11-13 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Urinary Incontinence; Quality of Life; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Urinary Incontinence; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bladder Training (Experimental): Patients in the structured bladder training group were trained on "lifestyle changes (nutrition, fluid management, exercise), pelvic floor muscle exercises and bladder control techniques".
  Interventions: Behavioral: Bladder Training
- Control Group (No Intervention): Routine patient training was given to the patients in the control group by a nurse working in the clinic.

INTERVENTIONS:
Behavioral: Bladder Training — Patients in the structured bladder training group were trained on "lifestyle changes (nutrition, fluid management, exercise), pelvic floor muscle exercises and bladder control techniques".
  Arms: Bladder Training

SUMMARY:
Radical prostatectomy is the gold standard in the treatment of patients with localized prostate cancer. Urinary incontinence, which is common after surgery, can affect the quality of life of men negatively. There are various attempts to prevent and treat urinary symptoms after radical prostatectomy.The aim of this study is to evaluate the effect of the structured bladder training program on lower urinary tract symptoms and quality of life in patients undergoing radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 40 years
* Being male
* Being with localized prostate cancer
* Undergoing open radical prostatectomy
* No preoperative urinary incontinence
* Being body mass index> 30 kg/m2
* Agreeing to participate in the research
* Being literate

Exclusion Criteria:

* Having a congenital disorder of the urinary system
* Having neurological disorders
* Having a history of transurethral resection of the prostate
* Having communication and mental impairment
* Inability to do pelvic floor muscle exercises

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-11-07 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence-related quality of life assessed by the International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) | 3 months after from baseline (0 month)
  The primary endpoint of this study was the difference between groups in terms of International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) scores 3 months after. This scale consists of 6 questions.The range of scores obtained from the scale varies between 0-21 points. High scores on the scale indicate that the quality of urinary incontinence is severely affected.

SECONDARY OUTCOMES:
Lower urinary tract symptoms assessed by the International Consultation on Incontinence Questionnaire-Male Lower Urinary Tract Symptoms (ICIQ-MLUTS) | 3 months after from baseline (0 month)
  The secondary endpoint is the difference between the groups in terms of International Consultation on Incontinence Questionnaire-Male Lower Urinary Tract Symptoms (ICIQ-MLUTS) scores after 3 months. This scale consists of 13 questions. Each question has a 4-point severity scale (0-4) and a 10-point visual analog scale (0-10) measuring quality of life. As the scores obtained from the scale increase, complaints about urinary system symptoms increase and the quality is negatively affected.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gezginci, RN, PhD, Principal Investigator — Saglik Bilimleri Üniversitesi
Locations (1):
- Elif Gezginci, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tienforti D, Sacco E, Marangi F, D'Addessi A, Racioppi M, Gulino G, Pinto F, Totaro A, D'Agostino D, Bassi P. Efficacy of an assisted low-intensity programme of perioperative pelvic floor muscle training in improving the recovery of continence after radical prostatectomy: a randomized controlled trial. BJU Int. 2012 Oct;110(7):1004-10. doi: 10.1111/j.1464-410X.2012.10948.x. Epub 2012 Feb 14. PMID 22332815
- [Background] Jarvis TR, Sandhu JS. Management of urinary incontinence after radical prostatectomy. Curr Urol Rep. 2014 Jul;15(7):421. doi: 10.1007/s11934-014-0421-6. PMID 24859671
- [Background] de Lira GHS, Fornari A, Cardoso LF, Aranchipe M, Kretiska C, Rhoden EL. Effects of perioperative pelvic floor muscle training on early recovery of urinary continence and erectile function in men undergoing radical prostatectomy: a randomized clinical trial. Int Braz J Urol. 2019 Nov-Dec;45(6):1196-1203. doi: 10.1590/S1677-5538.IBJU.2019.0238. PMID 31808408
- [Background] Hodges P, Stafford R, Coughlin GD, Kasza J, Ashton-Miller J, Cameron AP, Connelly L, Hall LM. Efficacy of a personalised pelvic floor muscle training programme on urinary incontinence after radical prostatectomy (MaTchUP): protocol for a randomised controlled trial. BMJ Open. 2019 May 5;9(5):e028288. doi: 10.1136/bmjopen-2018-028288. PMID 31061057
- [Background] Bernardes MFVG, Chagas SC, Izidoro LCR, Veloso DFM, Chianca TCM, Mata LRFPD. Impact of urinary incontinence on the quality of life of individuals undergoing radical prostatectomy. Rev Lat Am Enfermagem. 2019 Mar 10;27:e3131. doi: 10.1590/1518-8345.2757.3131. PMID 30916232
- [Background] Chang JI, Lam V, Patel MI. Preoperative Pelvic Floor Muscle Exercise and Postprostatectomy Incontinence: A Systematic Review and Meta-analysis. Eur Urol. 2016 Mar;69(3):460-7. doi: 10.1016/j.eururo.2015.11.004. Epub 2015 Nov 21. PMID 26610857